CLINICAL TRIAL: NCT02839889
Title: A Study to Assess the Tolerability, Safety, and Feasibility of Naloxegol in Patients With Cancer and Opioid-Induced Constipation
Brief Title: Tolerability, Safety, and Feasibility of Naloxegol in Patients With Cancer and OIC (Opioid Induced Constipation)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped due to challenges recruiting eligible patients.
Sponsor: Hospice of Henderson County, Inc. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Janet Bull, Chief Medical Officer, Hospice of Henderson County, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3820C00041
Record Dates: First submitted 2016-06-17; First posted 2016-07-21 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Cancer; Constipation; Pain
MeSH Terms: conditions — Neoplasms; Constipation; Pain | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo once daily for two weeks
  Interventions: Drug: Placebo
- Naloxegol (Active Comparator): Naloxegol 25mg tablets once daily for two weeks
  Interventions: Drug: Naloxegol

INTERVENTIONS:
Drug: Naloxegol — Naloxegol 25mg tablets for two weeks, followed by a two week open-label period
  Other Names: Movantik
  Arms: Naloxegol
Drug: Placebo — Placebo once daily for two weeks, followed by two week open-label period
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if naloxegol can be used in the treatment of opioid-induced constipation in patients with cancer and pain. This phase 4 study consists of a two week randomized double blind period followed by a two week open-label period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older: Women of child bearing potential must have a negative urine pregnancy test during the Screening/Opioid Induced Constipation (OIC) Confirmation/Baseline period, a history of no sexual activity or consistent use of an effective birth control method for at least 12 weeks prior to the study, and agreement that no sexual activity or the method of birth control will be continued during the study and for a period of 8 weeks after it ends; male patients who are sexually active must agree to use a barrier method of contraception (condom with spermicide) from the first dose of Investigational Product until 12 weeks after their last dose
* Able to follow instructions in English, give informed consent and to answer patient reported outcomes (PRO) questions by himself/herself; the patient will provide written informed consent before initiation of any study-related procedures
* Active cancer of any type with an investigator-estimated life expectancy ≥ 8 weeks and a Palliative Performance Status scale score ≥ 30%
* Patients receiving concurrent chemotherapy must have received and recovered from a minimum of 1 cycle of the current chemotherapy regimen upon consenting to the study and be considered stable in the opinion of the investigator
* Chronic cancer-related pain, defined as pain for a minimum of ≥2 weeks which on review by the investigator, can be attributed to the neoplasm or its treatment
* Daily treatment with an opioid drug which is taken at a dose equal to or greater than 20 mg morphine or its equivalent for at least one week, with no expectation of a decrease greater than 25% or an increase greater than 100% during the study period.
* Patients may or may not be on a stable laxative regimen, defined as daily use at a stable dose for >7 days; if the patient is taking a stable dose, he or she must be willing to remain on that regimen for the 7 day confirmation period without titration or adjustments.

History of constipation, defined through history and through participation in the Screening/OIC Confirmation/Baseline period:

* Patient history must include 2 or more of the following during defecations occurring in the two weeks prior to screening:
* <3 spontaneous bowel movements per week
* hard/lumpy stools (Bristol Stool Scale Type 1 or 2) in more than 25% of defecations
* sensation of incomplete evacuation in more than 25% of defecations
* sensation of anorectal obstruction in more than 25% of defecations
* Straining during more than 25% of defecations

Note: (spontaneous bowel movements (SBMs) are defined as not using a laxative if not already taking daily laxatives, or if taking daily laxatives, not using an additional laxative).

* Confirmation during the 7-day OIC confirmation period must include at least 2 or more of the following symptoms:
* <3 SBMs per week
* hard/lumpy stools (Bristol Stool Scale Type 1 or 2) in more than 25% of defecations
* sensation of incomplete evacuation in more than 25% of defecations
* sensation of anorectal obstruction in more than 25% of defecations
* Straining during more than 25% of defecations

Exclusion Criteria:

* Cancer-related/medical comorbidity-related

  * Patients with a past or current history of intra-abdominal neoplasm AND clinical findings that, on review by the investigator, may increase the risk of bowel perforation
  * An active condition associated with clinically significant brain pathology, including known brain metastases, meningeal metastases, past traumatic brain injury, multiple sclerosis, uncontrolled epilepsy with signs or symptoms of compromised blood brain barrier
  * Patients expected to undergo a first course of a chemotherapy regimen during the study period, patients who received a vinca alkaloid within 2 months, patients who have any history of vinca-associated GI autonomic neuropathy and/or constipation, or patients receiving a chemotherapy regimen including a VEGF-inhibitor (e.g., bevacizumab, sorafenib).
  * Requiring radiation therapy between the diaphragm and pelvis 2 weeks prior to Visit 1 (screening) and/or during the study
  * Any other significant and/or progressive condition (medical, neurological, psychiatric or metabolic) or symptom that could increase the risk of participation in the study or affect the interpretation of study data as determined by the investigator (e.g., uncontrolled hypothyroidism, inadequately controlled clinical depression, poorly controlled seizure disorder)
  * Hemorrhagic diathesis
  * Expected to have a surgical procedure requiring general anesthesia during the study period
* Other gastrointestinal disorders

  * Medical conditions and treatments, which in the judgment of the investigator, may be associated with diarrhea, intermittent loose stools, or constipation, (e.g., active diverticular disease, peritonitis of any cause, inflammatory bowel disease, active irritable bowel syndrome, chronic idiopathic constipation).
  * Any conditions that could affect the absorption or metabolism of the study drug (e.g., malabsorption syndrome, severe liver disease) as judged by the investigator
  * Evidence of fecal impaction either by physical or x-ray exam
  * Known or suspected mechanical GI obstruction
  * Current peritoneal catheter for intra-peritoneal chemotherapy or dialysis
  * Fecal ostomy
  * History of fecal incontinence
  * History of bowel surgery within 60 days of the screening period
  * Any other potential non-opioid cause of bowel dysfunction that in opinion of investigator might be a contributor to the constipation
* Pain-related

  * Receiving opioid medication on less than daily dosing schedule only
  * Severe background pain (eg, typical average daily pain intensity rating of 8 to 10 on an 11-point NRS) refractory opioid therapy
* Any of the following findings or conditions between the enrollment and randomization visits:

  * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x upper limit normal (ULN) and/or serum bilirubin >2 x ULN (unless elevation is due to Gilbert's syndrome)
  * Calculated Creatinine clearance <30 ml/min
  * A Fridericia corrected QT interval (QTcF) > 500 msec at screening, history of myocardial infarction within 6 months before randomization, symptomatic congestive heart failure despite treatment, unstable angina, or symptomatic peripheral vascular disease
  * Active substance or alcohol use that, in the opinion of the investigator, may compromise patient's ability to comply with the study instructions
  * Use of prohibited medications as listed in Section 5.5
  * Pregnancy or lactation
  * Known history of intolerance or hypersensitivity to alvimopan, methylnaltrexone, or other peripherally acting opioid antagonists or to any other component in the tablets
  * Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff, staff at the study site, and third-party vendors)
  * Any receipt of an investigational medication within 30 days of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09; Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Bull, MD, Principal Investigator — Hospice of Henderson County, Inc.
Locations (3):
- United States (3):
  - MJHS Institute for Innovation in Palliative Care, New York, New York
  - Hospice of Henderson County, Inc, Flat Rock, North Carolina
  - Hospice of the Western Reserve, Inc., Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multi center was conducted at 3 sites in the US. Enrollment to the study was stopped due to recruitment challenges and no new patients have been screened as of January 2018. 5 patients were randomized across the 2 treatment groups.
Pre-assignment Details: To confirm eligibility participants underwent a 7 day baseline assessment/OIC confirmation period. 12 patients provided consent for this study, however 7 did not fulfill eligibility criteria during the 7 day baseline period.
Period: Randomization Period
Arm/Group | Placebo | Naloxegol
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0
Period: Open-Label Period
Arm/Group | Placebo | Naloxegol
Started | 0 | 5
Completed | 0 | 4
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Naloxegol | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5
Baseline Numerical Rating Scale (NRS) for Pain [Mean (Full Range); unit: score on a scale] — Baseline Numerical Rating Scale (NRS) for Pain during the OIC Confirmation Period. Numeric Rating Scale is 0-10. 0 is no pain and 10 is worst possible pain. Lower values are a better outcome and higher values are a worse outcome.
  score on a scale | 5.7 [5.1 to 6.3] | 6.2 [5.4 to 7.1] | 6.0 [5.1 to 7.1]
Baseline Electrocardiogram QTC Interval [Mean (Full Range); unit: Milliseconds] | 430.8 [423 to 438.5] | 414.5 [381.6 to 447] | 421 [381.6 to 447]
Baseline Electrocardiogram Heart Rate [Mean (Full Range); unit: beats per minute] | 82 [80 to 84] | 79 [66 to 98] | 80.2 [66 to 98]
Baseline Daily Opioid Use [Mean (Full Range); unit: morphine milligram equivalents per day] | 300 [240 to 360] | 126.5 [40 to 300] | 196 [40 to 360]
Baseline Systolic Blood Pressure [Mean (Full Range); unit: mmHg] | 133.5 [110 to 157] | 118 [88 to 150] | 124.2 [88 to 157]
Baseline Diastolic Blood Pressure [Mean (Full Range); unit: mmHg] | 85 [76 to 94] | 71.3 [56 to 96] | 76.8 [56 to 96]
Baseline Pulse Rate [Mean (Full Range); unit: beats per minute] | 81 [78 to 84] | 79 [60 to 104] | 79.8 [60 to 104]
Baseline Bristol Stool Scale score [Mean (Full Range); unit: score on a scale] — The Bristol Stool Scale classifies the type of bowel movement on a scale from 1-7, based on the appearance of stool. 1 indicates severe constipation, 2 indicates mild constipation, 3-4 indicate a normal bowel movement, 5 indicates that the patient is lacking dietary fiber, 6 indicates mild diarrhea, and 7 indicates severe diarrhea. A better score would trend toward the middle of the scale (ranges 3-4), while scores at either end of the scale correspond to worse outcomes.
  score on a scale | 3.91 [2.17 to 5.64] | 1.94 [1.75 to 2.33] | 2.73 [1.75 to 5.64]
Baseline Respiratory Rate [Mean (Full Range); unit: breaths per minute] | 14 [12 to 16] | 15.3 [12 to 20] | 14.8 [12 to 20]
Baseline Degree of Straining [Mean (Full Range); unit: score on a scale] — Degree of straining scale measures the amount of straining during a bowel movement. The scale is 1 to 5 with 1 being "not at all" and 5 being "an extreme amount". Lower scores are better and higher scores are worse.
  score on a scale | 2.21 [1.91 to 2.5] | 2.06 [1.17 to 3.25] | 2.12 [1.17 to 3.25]
Baseline Complete Evacuation with Bowel Movements [Mean (Full Range); unit: % of days with complete evacuation] | 39.3 [28.6 to 50] | 41.7 [25 to 62.5] | 40.7 [25 to 62.5]
Baseline Patient Assessment of Constipation Symptom Assessments (PAC-SYM) [Mean (Full Range); unit: score on a scale] — The PAC-SYM is divided into three subscales. Each item is scored 0-4. Items 1-4 measure abdominal symptoms (total subscale range 0-16), items 5-7 measure rectal symptoms (total subscale score 0-12), and items 8-12 measure stool symptoms (total subscale range 0-20). For each subscale, lower scores are better and higher scores are worse.
  The total construct score is generated by summing the scores of the subscales. This total score ranges from 0-48, with lower scores corresponding to better outcomes, and higher scores corresponding to worse outcomes.
  score on a scale
    Abdominal symptoms | 6.5 [5 to 8] | 8 [7 to 9] | 7.4 [5 to 9]
    Rectal Symptoms | 2 [1 to 3] | 3.3 [2 to 4] | 2.8 [1 to 4]
    Stool symptoms | 7.5 [6 to 9] | 8 [3 to 15] | 7.8 [3 to 15]
    Total Score | 16 [12 to 20] | 19.3 [13 to 28] | 18 [12 to 28]
Baseline Patient Assessment of Constipation (PAC-QOL) [Mean (Full Range); unit: score on a scale] — The PAC-QOL is a 28-item questionnaire divided into 4 subscales. Each item is scored 0-4. Items 1-4 measure physical discomfort (total subscale range 0-16), 5-12 measure psychosocial discomfort (range 0-32), 13-23 measure worries/concerns (range 0-44), and 24-28 measure satisfaction (range 0-20). For each subscale, lower scores are better and higher scores are worse.
  The total score is generated by summing the scores of the subscales. This total score ranges from 0-112, with lower scores corresponding to better outcomes, and higher scores corresponding to worse outcomes.
  score on a scale
    Physical Discomfort | 8 [7 to 9] | 4.7 [2 to 10] | 6 [2 to 10]
    Psychosocial discomfort | 14 [6 to 22] | 4.3 [0 to 9] | 8.2 [0 to 22]
    Worries/concerns | 17 [11 to 23] | 15.3 [8 to 25] | 16 [8 to 25]
    Satisfaction | 5.5 [5 to 6] | 3.3 [2 to 5] | 4.2 [2 to 6]
    Total Score | 44.5 [31 to 58] | 27.7 [13 to 46] | 34.4 [13 to 58]

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) for Pain Change From Baseline
Description: Change from baseline in mean daily NRS (Numerical Rating Scale) values will be calculated as the post-baseline value minus the baseline. Baseline NRS is the mean daily NRS values recorded during the Opioid Induced Constipation (OIC) Confirmation period. Numeric Rating Scale is 0-10. 0 is no pain and 10 is worst possible pain. Lower values are a better outcome and higher values are a worse outcome. Post-baseline values were calculated as the mean of NRS scores during visits 2-4.
Time Frame: Assessed from screening/Opioid Induced Constipation (OIC) Confirmation period through study completion, approximately 6 weeks.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
score on a scale | 0.65 [0.3 to 1] | .33 [-0.4 to 1.4]

2. Primary Outcome: Daily Opioid Use Change From Baseline
Description: Change from baseline in mean daily opioid dose will be calculated as the post-baseline value minus the baseline value. Positive changes from baseline indicate there was a need to increase the opioid dose. Baseline daily opioid dose is the mean daily opioid dose recorded during the Opioid Induced Constipation (OIC) Confirmation period.
Time Frame: Assessed from screening through study completion, approximately 6 weeks.
Measure: Mean (Full Range); unit: morphine milligram equivalents per day
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
morphine milligram equivalents per day | 1144 [0 to 2288] | 20 [0 to 60]

3. Primary Outcome: Adverse Events Associated With Blood Laboratory Result Changes From Baseline
Description: Changes from Baseline to Visit 3 (approximately Day 15) for all patients will be calculated as the post-baseline test value minus the baseline test value.
Time Frame: Change from Baseline at End of Double Blind Phase (Visit 3, approximately day 15)
Population: All abnormal lab values were deemed not clinically significant by Investigators. Therefore, changes did not meet the criteria for an adverse event and changes were not collected.
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Electrocardiogram QTC Interval
Description: Changes from Baseline to Visit 3 (approximately Day 15) for Electrocardiogram (ECG) QTC interval data will be derived by subtracting the baseline value from the final assessment data.
Time Frame: Change from Baseline at End of Double Blind Phase (Visit 3, approximately day 15)
Measure: Mean (Full Range); unit: milliseconds
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
milliseconds | -24.8 [-61.6 to 12] | -6.9 [-17 to 4]

5. Primary Outcome: Electrocardiogram Heart Rate
Description: Changes from Baseline to Visit 3 (approximately Day 15) for Electrocardiogram (ECG) heart rate data will be derived by subtracting the baseline value from the final assessment data.
Time Frame: Change from Baseline at End of Double Blind Phase (Visit 3, approximately day 15)
Measure: Mean (Full Range); unit: beats per minute
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
beats per minute | 9 [7 to 11] | 10 [2 to 23]

6. Primary Outcome: Change From Baseline in Systolic Blood Pressure
Description: Change from Baseline in systolic blood pressure at post baseline (visits 2, 3, 4) will be derived as the value at the visit minus the baseline value for the same assessment. The post-baseline values were calculated as a mean of values from visits 2 through 4.
Time Frame: Change from Baseline in systolic blood pressure through study completion, approximately 6 weeks.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
mmHg | -10.3 [-30.3 to 9.7] | -8.8 [-19 to 7.3]

7. Primary Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Change from Baseline in diastolic blood pressure at post baseline (visits 2, 3, 4) will be derived as the value at the visit minus the baseline value for the same assessment. The post-baseline values were calculated as a mean of values from visits 2 through 4.
Time Frame: Change from Baseline in diastolic blood pressure through study completion, approximately 6 weeks.
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
mmHg | -10.5 [-20 to -1] | -1.8 [-9.3 to 4]

8. Primary Outcome: Change From Baseline in Respiratory Rate
Description: Change from Baseline in respiratory rate at post baseline (visits 2, 3, 4) will be derived as the value at the visit minus the baseline value for the same assessment. The post-baseline values were calculated as a mean of values from visits 2 through 4.
Time Frame: Change from Baseline in respiratory rate through study completion, approximately 6 weeks.
Measure: Mean (Full Range); unit: breaths per minute
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
breaths per minute | 1.7 [-2 to 5.3] | 1.2 [-0.7 to 3.7]

9. Primary Outcome: Change From Baseline in Pulse Rate
Description: Change from Baseline in pulse rate at post baseline (visits 2, 3, 4) will be derived as the value at the visit minus the baseline value for the same assessment. The post-baseline values were calculated as a mean of values from visits 2 through 4.
Time Frame: Change from Baseline in pulse rate through study completion, approximately 6 weeks.
Measure: Mean (Full Range); unit: beats per minute
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
beats per minute | 4.5 [3.7 to 5.3] | 10.3 [5.3 to 15.3]

10. Secondary Outcome: Rescue Free Bowel Movements (RFBM) Responder Rate
Description: Daily diary data will be used to identify RFBMs. The weekly RFBM frequency within each time period will be calculated as: (Total number of RFBMs during the time period of interest/number of days) x 7. RFBM rate calculated from post baseline period.
Time Frame: Assessed from Baseline through Study Completion, approximately 6 weeks.
Measure: Mean (Full Range); unit: RFBMs/days *7
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
RFBMs/days *7 | 8.14 [3.5 to 12.79] | 3.82 [1.59 to 5.55]

11. Secondary Outcome: Time to First Post-dose Rescue Free Laxation
Description: Time (in hours) to first post-dose rescue free bowel movement minus first dose date and time.
Time Frame: First dose date to first post-dose rescue free bowel movement
Measure: Mean (Full Range); unit: Hours
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
Hours | 23.3 [17.96 to 28.58] | 33.5 [3.67 to 67.73]

12. Secondary Outcome: Bristol Stool Scale (BSS) Score
Description: The Bristol Stool Scale classifies the type of bowel movement on a scale from 1-7, based on the appearance of stool. 1 indicates severe constipation, 2 indicates mild constipation, 3-4 indicate a normal bowel movement, 5 indicates that the patient is lacking dietary fiber, 6 indicates mild diarrhea, and 7 indicates severe diarrhea. A better score would trend toward the middle of the scale (ranges 3-4), while scores at either end of the scale correspond to worse outcomes.
  Bristol Stool Scale (BSS) Score calculated by the sum of daily BSS scores divided by the number of bowel movements that occurred from baseline to study completion. Change from Baseline calculated as the Baseline value minus the post-baseline value.
Time Frame: Assessed from baseline through Study Completion, approximately 6 weeks.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
score on a scale | -.06 [-.4 to .28] | 2.37 [1.51 to 3.02]

13. Secondary Outcome: Patient Assessment of Constipation Symptoms (PAC-SYM)
Description: The PAC-SYM is divided into three subscales. Each item is scored 0-4. Items 1-4 measure abdominal symptoms (total subscale range 0-16), items 5-7 measure rectal symptoms (total subscale score 0-12), and items 8-12 measure stool symptoms (total subscale range 0-20). For each subscale, lower scores are better and higher scores are worse.
  The total construct score is generated by summing the scores of the subscales. This total score ranges from 0-48, with lower scores corresponding to better outcomes, and higher scores corresponding to worse outcomes.
  Change from baseline in mean values calculated as post-baseline value minus baseline value for each scale, and for total. Post-baseline values defined as the mean of day 15 and day 29.
Time Frame: day 1, day 15, day 29
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
score on a scale
  Abdominal Symptoms | 1 [0 to 2] | .5 [-2 to 3]
  Rectal Symptoms | 1.25 [1 to 1.5] | 1.2 [-1.5 to 5]
  Stool Symptoms | .5 [-0.5 to 1.5] | -.2 [-1.5 to 1.5]
  Total Score | 2.75 [2.5 to 3] | 1.5 [-3.5 to 9.5]

14. Secondary Outcome: Patient Assessment of Constipation Quality of Life (PAC-QOL)
Description: The PAC-QOL is a 28-item questionnaire divided into 4 subscales. Items 1-4 measure physical discomfort (subscale range 0-16), 5-12 measure psychosocial discomfort (range 0-32), 13-23 measure worries/concerns (range 0-44), and 24-28 measure satisfaction (range 0-20). For each subscale, lower scores are better and higher scores are worse.
  The total score is generated by summing the scores of the subscales. This total score ranges from 0-112, with lower scores corresponding to better outcomes, and higher scores corresponding to worse outcomes.
  Change from baseline in mean values calculated as post-baseline value minus baseline value for each subscale, and for total. Post-baseline values defined as the mean of day 15 and day 29.
Time Frame: day 1, day 15, day 29
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
score on a scale
  Physical discomfort | -1.25 [-1.5 to -1] | 0.17 [0 to 0.5]
  Psychosocial Discomfort | -1 [-9 to 7] | 6 [1 to 14]
  Worries/concerns | 1.5 [-3.5 to 6.5] | 1.17 [-1.5 to 3.5]
  Satisfaction | 3.5 [2 to 5] | 3.83 [2 to 6.5]
  Total Score | 2.75 [-12 to 17.5] | 11.17 [5.5 to 20]

15. Secondary Outcome: Degree of Straining Question With Each Bowel Movement
Description: Degree of straining scale is 1 to 5 with 1 being "not at all" and 5 being "an extreme amount". Lower scores are better and higher scores are worse.
  Change from baseline in mean values calculated as the post baseline value minus the baseline. Degree of Straining scale change from baseline mean scores calculated from baseline to study completion.
Time Frame: Assessed at baseline through Study Completion with each bowel movement, approximately 6 weeks.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
score on a scale | .6 [-.31 to 1.5] | -.35 [-.67 to .09]

16. Secondary Outcome: Complete Evacuation Question With Each Bowel Movement
Description: Change from Baseline in mean values calculated as the post baseline value minus the baseline. The post baseline value is the percentage of days from baseline to study completion with at least one complete bowel evacuation.
Time Frame: Assessed at baseline through Study Completion with each bowel movement, approximately 6 weeks.
Measure: Mean (Full Range); unit: % of days with complete evacuation
Arm/Group | Placebo | Naloxegol
Number analyzed (Participants) | 2 | 3
% of days with complete evacuation | 21.92 [21.43 to 22.41] | 7.7 [-11.36 to 79.31]

ADVERSE EVENTS:
Time Frame: Occurrences from Baseline through study completion, approximately 6 weeks
Arm/Group | Placebo | Naloxegol
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | Naloxegol (N=3)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
fever (General disorders) | 1 (1) | 0 (0)
chills (General disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
abdominal distention (General disorders) | 1 (1) | 0 (0)
bladder spasms (Renal and urinary disorders) | 0 (0) | 1 (1)
increased back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
increased abdominal pain (General disorders) | 0 (0) | 1 (1)
worsening constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
mental status changes (Nervous system disorders) | 0 (0) | 1 (1)
abdominal cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to significant recruitment challenges enrollment was stopped. Only 5 patients were randomized (less than 12% of expected). There was insufficient data to perform the protocol specified analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT02839889/Prot_SAP_000.pdf